CLINICAL TRIAL: NCT03100968
Title: Utility of Ultrasound in Identification of Midline and Placement of Epidural in Severely Obese Parturients: A Randomized, Prospective Study
Brief Title: Utility of Ultrasound in Identification of Midline and Placement of Epidural in Severely Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mark Powell, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F150402002
Record Dates: First submitted 2017-03-25; First posted 2017-04-04 (Actual); Results first posted 2019-09-17 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Epidural Anesthesia; Spinal Ultrasound; Obesity
MeSH Terms: conditions — Obesity | interventions — Ultrasonography

STUDY DESIGN:
Intervention Model Description: Upon enrollment into the study, participants will be randomized 1:1 to either ultrasound or palpation. Randomization will be performed via random drawing: the provider will randomly select a card assigning the method of midline identification (i.e., ultrasound or palpation). Anesthesia providers will not be randomized. Any qualified provider available to place the epidural will be the person to perform the procedure.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Palpation Group (Active Comparator): The palpation group will have an epidural placed after manual palpation of the spine.
  Interventions: Procedure: Palpation
- Ultrasound Group (Active Comparator): The ultrasound group will have an epidural placed after identifying midline with the ultrasound.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Procedure: Palpation — Traditional epidural methods used for the identification of the midline using palpation prior to procedure
  Arms: Palpation Group
Device: Ultrasound — Lumbar spinal ultrasound performed for identification of the midline prior to procedure.
  Arms: Ultrasound Group

SUMMARY:
This study will address the utility of ultrasound in the placement of an epidural catheter in severely obese parturients. Identification of midline can often be difficult using the standard method of palpation in obese patients. The Investigator will determine if the use of ultrasound decreases the amount of time and number of attempts required to place the epidural.

DETAILED DESCRIPTION:
The use of ultrasound has expanded into many areas of medicine including the identification of bony landmarks to facilitate epidural placement in obstetric anesthesia. Using ultrasound for epidural placement has become popular over the last decade with several studies being published on the topic. The likely increase in popularity for ultrasound use in the obstetric population is the need to more reliably locate bony landmarks as the traditional palpation technique has been shown to be an inaccurate way to accomplish this. Given the fact that the long-taught palpation technique can be inaccurate and studies have validated the use of ultrasound for epidural placement, ultrasound technique is routinely taught by the obstetric anesthesiologists to the anesthesiology residents at the University of Alabama at Birmingham (UAB). Also, since both techniques are considered standard practice at UAB, anesthesia providers (residents, fellows, and faculty) are free to choose either technique to locate bony structures of the back prior to epidural placement. Since no current study has specifically addressed its use in the obese pregnant patient, the investigators would like to validate its use in this population.

In this study, investigators will evaluate the use of ultrasound in the obese population to determine if its use will decrease the time it takes to place the epidural and number of attempts required when compared to the traditional palpation technique. The study will also determine the success rate of epidural placement in both the palpation and ultrasound groups.

ELIGIBILITY:
Inclusion Criteria:

* patient request for a labor epidural
* BMI≥35

Exclusion Criteria:

* BMI<35
* patient refusal of a labor epidural
* coagulopathy
* platelets<80,000
* prior spine procedure or instrumentation
* a diagnosis of scoliosis
* an intracranial or spinal mass

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All female parturients in active labor
Enrollment: 150 (Actual)
Dates: Start 2015-06-22 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F Powell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Palpation Group | Ultrasound Group
Started | 75 | 75
Completed | 75 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Palpation Group | Ultrasound Group | Total
Number analyzed (Participants) | 75 | 75 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 75 | 150
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 75 | 150
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 75 | 75 | 150
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 44.4 (6.9) | 43.3 (7.1) | 43.8 (7.0)
Height [Mean (Standard Deviation); unit: Centimeters] | 163.9 (8.2) | 164.2 (7.1) | 164.1 (7.7)
Weight [Mean (Standard Deviation); unit: Kilograms] | 119.5 (20.6) | 116.8 (20.2) | 118.1 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Time for Epidural Placement
Description: Comparing the time it takes for epidural placement in the palpation group vs. the ultrasound group. Measured in minutes from local anesthesia skin wheal to administration of the epidural test dose.
Time Frame: Baseline up to 1 hour
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
minutes | 9.0 (6.8) | 6.2 (3.8)

2. Primary Outcome: Number of Needle Passes
Time Frame: Baseline up to 1 hour
Measure: Mean (Standard Deviation); unit: needle passes
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
needle passes | 2.8 (2.0) | 2.1 (1.4)

3. Primary Outcome: Total Time
Time Frame: Baseline up to 1 hour
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
Minutes | 9.5 (6.8) | 6.9 (3.9)

4. Secondary Outcome: Time to Identify Midline
Description: Comparing the time it takes to locate midline of the back in the palpation group vs. the ultrasound group. Measured in minutes from the start of the identification process until completion of the midline identification process.
Time Frame: Baseline up to 1 hour
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
seconds | 30.9 (16.3) | 44.5 (24.7)

5. Secondary Outcome: Epidural Failure Rate
Description: Comparing the number of epidural failures in the palpation vs. ultrasound group.
Time Frame: Baseline up to 1 hour
Measure: Number; unit: failed epidurals
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
failed epidurals | 7 | 3

6. Secondary Outcome: Number of Top-offs Required
Time Frame: Baseline up to 1 hour
Measure: Mean (Standard Deviation); unit: number of topoffs required
Arm/Group | Palpation Group | Ultrasound Group
Number analyzed (Participants) | 75 | 75
number of topoffs required | 0.5 (1.1) | 0.4 (0.9)

ADVERSE EVENTS:
Time Frame: Baseline up to 1 hour
Arm/Group | Palpation Group | Ultrasound Group
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/75
Other Adverse Events (participants affected / at risk) | 0/75 | 0/75

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT03100968/Prot_SAP_000.pdf